CLINICAL TRIAL: NCT02555163
Title: Holmium (Ho: YAG) Laser En Bloc Resection Of Bladder Tumor (HoLERBT) Versus Conventional Transurethral Resection Of Bladder Tumors (cTURBT): A Prospective Randomized Controlled Trial
Brief Title: Laser En Bloc Resection Of Bladder Tumor (HoLERBT) VS. Conventional Transurethral Resection Of Bladder Tumors (cTURBT)
Acronym: HoLERBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Elshal, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD.15.165.
Record Dates: First submitted 2015-09-16; First posted 2015-09-21 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Bladder Cancer
Keywords: bladder cancer, laser
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HoLERBT (Experimental): Holmium (Ho: YAG) Laser En Bloc Resection Of Bladder Tumor
  Interventions: Device: HoLERBT
- cTURBT (Active Comparator): Conventional Transurethral Resection Of Bladder Tumors
  Interventions: Device: cTURBT

INTERVENTIONS:
Device: HoLERBT — Using holmium laser, the tumour will be removed as one piece from its base working underneath the muscle layer
  Arms: HoLERBT
Device: cTURBT — using the conventional electrocautery device with the cutting hot loop the tumor will be removed in pieces
  Arms: cTURBT

SUMMARY:
Randomized clinical trial aiming to assess Holmium Laser En Bloc Resection Of Bladder Tumor (HoLERBT) in comparison with Conventional Transurethral Resection Of Bladder Tumors (cTURBT) in tumor histopathological staging quality, detrusor muscle sampling in biopsy, completeness of tumor resection and peri procedure complication.

DETAILED DESCRIPTION:
Urothelial carcinoma of the bladder is the 2nd most common urological malignancy and it makes a growing healthcare problem worldwide.

The vast majority of newly diagnosed are non-muscle bladder cancers (NMIBC) which represents about 75% and can be treated with transurethral resection of bladder tumors (TURBT) so, correct initial staging is critical. The quality of TURBT strongly determines patient prognosis and overall treatment.

Conventional transurethral resection of bladder tumors (cTURBT) causes fragmentation, artifacts, thermal damages and tangential sections that might hamper histopathological evaluation.

The expert meeting at Davos of the European Association of Urology (EAU) section of Uro-Technology (ESUT) and the section of Uro-Oncology (ESOU) identified en bloc resections of bladder tumors (ERBT) using various energy sources or modified resection loops as a promising technique.

Laser therapy for the treatment of non muscle invasive bladder tumor (NMIBC) was first reported in the 1970s. Neodymium:YAG lasers were mainly used for tissue vaporization. Afterward, the introductions of en bloc resection methods have laser treatments for bladder cancer regains its popularity. The most commonly used are holmium (Ho:YAG) and thulium (Tm:YAG).

EBRBT overall complication rate of 0.7%, of which all complications had not been life-threatening. Compared conventional TURBT to HoLERBT, a significant reduction of obturator nerve reflex, related bladder perforations, peri- or postoperative bleeding was rare, reduction in bladder irrigation time in comparison with conventional TURB. Better histopathological results were with laser en bloc resection of bladder cancer by lowering of thermal damage The study will be conducted in a single tertiary centre at Urology and Nephrology Center in Mansoura, Egypt.

Eligible patient presented with papillary bladder tumor will be asked to participate in this study and will be provided with an informed consent form in line with Good Clinical Practise and the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed at the out-patient cystoscopy with papillary bladder tumour will be legible for inclusion

Exclusion Criteria:

* Tumor criteria

  * Non papillary gross features of the tumor
  * Anteriorly located tumor
* Patients criteria
* Poor performance status
* History of BCG sepsis
* History of bladder irradiation
* Contracted bladder

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
residual disease at re-staging transurethral bladder biopsy | 4 weeks after primary procedure
  Rebiopsy of the tumor base for detection of any residual disease at re staging TUR 4 weeks after primary procedure. Number of patients with residual disease at restaginf TUR will be counted in each arm and compared

SECONDARY OUTCOMES:
periprocedure complications | 2 days
  Modified Clavien scale will be used for reporting and comparison of periprocedure complications
recurrence free survival | 1 year
  Number of patients surviving for one year without tumor recurrence will be counted and compared

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Elshal, MD, Study Director — Mansoura urology and nephrology center, Mansoura University, Egypt
Locations (1):
- Urology and Nprhology Center, Al Mansurah, Aldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hashem A, Mosbah A, El-Tabey NA, Laymon M, Ibrahiem EH, Elhamid MA, Elshal AM. Holmium Laser En-bloc Resection Versus Conventional Transurethral Resection of Bladder Tumors for Treatment of Non-muscle-invasive Bladder Cancer: A Randomized Clinical Trial. Eur Urol Focus. 2021 Sep;7(5):1035-1043. doi: 10.1016/j.euf.2020.12.003. Epub 2020 Dec 30. PMID 33386289